CLINICAL TRIAL: NCT04639336
Title: Cognitive and Neurological Pathologies in Pompe Disease
Acronym: CNS
Status: Recruiting | Type: Observational
Sponsor: Duke University (Other)
Collaborators: Sanofi (Industry)
Responsible Party: Sponsor
Other Study IDs: Pro00072329
Record Dates: First submitted 2020-11-06; First posted 2020-11-20 (Actual); Last update posted 2025-04-17 (Actual); Status verified 2025-03

CONDITIONS: Pompe Disease
MeSH Terms: conditions — Glycogen Storage Disease Type II

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with Pompe disease

SUMMARY:
The purpose of this study is to better understand the long-term health effects of Pompe disease and to determine if there are any abnormal changes in the brain and peripheral nerves. Additionally, the investigators will study the relationship between the abnormal changes in brain, nervous system findings, and developmental outcomes.

The investigators will collect clinical information from clinic visits as well as assessments such as neuroimaging (magnetic resonance imaging (MRI), magnetic resonance spectroscopy (MRS), and diffusion tensor imaging (DTI)), cognition, academic skills, speech and language function, physical therapy and quantitative muscle ultrasound. Subjects will be in this study for at least 3 years and up to 6 years.

ELIGIBILITY:
Inclusion Criteria:

* Subject has a confirmed and documented diagnosis of infantile Pompe Disease (IPD) or Late onset Pompe Disease (LOPD)

Exclusion Criteria:

* Refusal to give informed consent

Ages: 0 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children with infantile Pompe disease. Children with late-onset Pompe disease
Sampling Method: Non-Probability Sample
Enrollment: 45 (Estimated)
Dates: Start 2016-08-03 (Actual); Primary Completion 2028-03 (Estimated); Study Completion 2029-03 (Estimated)

PRIMARY OUTCOMES:
To determine the involvement of central nervous system (CNS) pathology in long-term survivors of IPD and early diagnosed LOPD patients being treated with enzyme replacement therapy (ERT) as measure by neuroimaging. | up to 6 years

SECONDARY OUTCOMES:
To further investigate developmental outcomes, such as cognition, language, academic skills and fine motor skills, of children with Pompe disease as reported by patient performance report measures. | up to 6 years
To further investigate developmental outcomes, such as cognition, language, academic skills and fine motor skills, of children with Pompe disease as reported by parent report measures. | up to 6 years
To characterize the motor speech function in children with IPD and LOPD as reported auditory-perceptual and instrumental methods. | up to 6 years
To investigate the relationship between neuroimaging findings and developmental outcomes, over time, for children with Pompe disease, as reported by . | up to 6 years
To investigate the extent of muscle pathology, especially myopathy and neuropathy in the distal lower extremities, using screening questionnaires. | up to 6 years
To investigate the extent of muscle pathology, especially myopathy and neuropathy in the distal lower extremities, using quantitative muscle ultrasound. | up to 6 years

CONTACTS AND LOCATIONS:
Overall Officials: Priya Kishnani, MD, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Crisp KD, Neel AT, Amarasekara S, Marcus J, Nichting G, Korlimarla A, Kishnani PS, Jones HN. Assessment of Dysphonia in Children with Pompe Disease Using Auditory-Perceptual and Acoustic/Physiologic Methods. J Clin Med. 2021 Aug 16;10(16):3617. doi: 10.3390/jcm10163617. PMID 34441913
- [Result] Korlimarla A, Spiridigliozzi GA, Crisp K, Herbert M, Chen S, Malinzak M, Stefanescu M, Austin SL, Cope H, Zimmerman K, Jones H, Provenzale JM, Kishnani PS. Novel approaches to quantify CNS involvement in children with Pompe disease. Neurology. 2020 Aug 11;95(6):e718-e732. doi: 10.1212/WNL.0000000000009979. Epub 2020 Jun 9. PMID 32518148
- [Result] Korlimarla A, Spiridigliozzi GA, Stefanescu M, Austin SL, Kishnani PS. Behavioral, social and school functioning in children with Pompe disease. Mol Genet Metab Rep. 2020 Aug 5;25:100635. doi: 10.1016/j.ymgmr.2020.100635. eCollection 2020 Dec. PMID 32793419